CLINICAL TRIAL: NCT05654337
Title: Obesity Pathway Intervention Among Overweight and Obese Adults at Primary Care Centers in Hail, Saudi Arabia: A Randomized Clustered Trial
Brief Title: Obesity Pathway Intervention Among Overweight and Obese Adults at Primary Care Centers in Hail, Saudi Arabia
Acronym: Telehealth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The New Model of Care, Hail Health Cluster (Other Government)
Collaborators: Health Holding Company, Hail Health Cluster, Saudi Arabia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Hail Health Cluster
Record Dates: First submitted 2022-12-07; First posted 2022-12-16 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Lifestyle-related Condition
MeSH Terms: conditions — Mental Disorders | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary and physical activity plan and advice on lifestyle change (Experimental): Dietary and physical activity schedules and instructed lifestyle change advice provided by a trained health coach and dietary education provided by a trained and licensed dietitian to the obese and overweight at the primary care centre.
  Interventions: Other: Expert health counseling
- Routine care for cases with obesity and overwieght (No Intervention): Adults with obesity and overweight attending routine primary care clinics

INTERVENTIONS:
Other: Expert health counseling — Expert advice on dietary education, lifestyle change, and physical exercise schedule
  Other Names: Dietary education, lifestyle change, and physical exercise schedule
  Arms: Dietary and physical activity plan and advice on lifestyle change

SUMMARY:
The goal of this pragmatic trial is to test the benefit of using dietary advice and health coaching for physical activities for obese and overweight in lowering body weight and making them lead a healthy lifestyle. The advice will be provided by an expert dietician and health coach at the primary health care. The main questions it aims to answer are:

To what extent does the obesity pathway among overweight and obese adults implemented at primary health care Clinics work well in lowering weight? To what extent do the use of dietary advice and coaching for physical activities for obese and overweight implemented at primary health care Clinics work well in achieving a positive lifestyle change? Participants will be asked to participate in the obesity pathway at primary care centres. An expert dietician and health coach will be used to provide a schedule for dietary control and coaching for physical activities.

Researchers will compare the change in body weight and lifestyle among overweight and obese adults in the intervention versus the control group at the primary care centre.

Adopting a healthy lifestyle, standard weight, healthy dietary habits, plus wise efforts to lowering your body weight is valuable. These need advice from an expert dietician and health coach to prevent the risk of contracting diabetes, heart disease, and cancer.

DETAILED DESCRIPTION:
Leadership and a multisectoral approach are the cornerstones in tackling the prevention of non-communicable diseases in Saudi Arabia. A focus should be on physical inactivity, tobacco, and unhealthy diet using effective and cost-effective interventions.

The last updated clinical practice guideline for the non-pharmacological management of overweight and obese Saudi adults strongly suggests lifestyle intervention rather than usual care alone, individualized counselling interventions rather than a generic educational pamphlet, physical activity rather than no physical activity, and physical activity in addition to diet rather than diet alone.

Many countries had implemented taxes on unprocessed sugar or sugar-added foods for reducing their consumption and preventing obesity and other adverse health events. however, no concrete evidence of the effectiveness of the intervention on the ground.

Mobile intervention technologies like pedometers or accelerometers with displays, activity trackers, smartphones, or tablets have a great effect in supporting sustainable health behaviour, increasing physical activity, and preventing the risk of chronic disease.

Research Questions:

1. To what extent does the obesity pathway intervention among overweight and obese adults implemented at primary health care clinics effective in achieving weight reduction?
2. To what extent does individualize nurse counselling such as dietary education and physical activity intervention among overweight and obese adults implemented at primary health care clinics effective in achieving a positive lifestyle change?

General objective:

To estimate the effectiveness of the obesity pathway intervention (individualized nurse counselling: dietary education and physical activity) at primary health care clinic in achieving weight reduction and positive lifestyle changes among overweight and obese adults.

Specific Objectives:

Aim 1: To compare the proportion of weight reduction among overweight and obese adults in the intervention versus the control group (routine care) at the Primary Health Care Clinic.

Aim 2: To compare the change in lifestyle among overweight and obese adults in the intervention versus the control group at the primary health care clinic.

Literature Review:

Planning an established clinic-based weight reduction program requires paying attention to different barriers to the retention of patients in the program.

Research Design and Methods:

This is a six months clustered randomized trial that will recruit adults who are obese and overweight to attend a primary health care clinic in Hail city.

Participants (P):

The participants will be adults who are obese and overweight of both genders attending the selected health centres. The participants are expected to be adults aged 18 years and above. Children and young adults will be excluded. In addition, severely ill patients, and patients with mental disorders will be excluded. The participants will be assessed at the start to collect the baseline data about Body Mass Index (BMI) to report eligible participants. At the end of the trial, a similar report on BMI will be obtained for each participant at three and six months after the beginning of the trial. A qualitative assessment report on lifestyle changes i.e. dietary habits and physical activities will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60 with proven obesity and overweight

Exclusion Criteria:

* severely ill or patient with other chronic health conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 440 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
The percentage of obese and overweight who lose 5% of their weight among participants. | 6 month from the start of the study
  The percentage of obese patients who lose 5% of their weight among participants in the intervention versus the control group (routine care) at the primary care clinic. This will be measured using a scoring checklist at the clinic and a self-based assessment card,
The percentage of patients who reduced their weight by 5%, and achieved more than 70 % adherence rate | 6 month from the start of the study
  The percentage of patients who reduced their weight by 5%, and achieved more than 70 % adherence rate to the provided schedule of dietary habits and physical activity in the intervention group vs. the control group

CONTACTS AND LOCATIONS:
Overall Officials: Meshari Aljamani, MOC Lead, Study Chair — Hail Health Cluster; Sultan N AlShammary, KSS Hospital Director, Study Director — New Model of Care, Hail Health Cluser; Mohammad S Altamimi, Data Quality Manager at HHC, Study Director — New Model of Care, Hail Health Cluster; Adel A Al Zuhair, Model of Care Project Manager, Study Director — New Model of Care, Hail Health Cluster
Locations (1):
- New Model of Care at Hail Health Cluster, Hail, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elfakki FA, Aljamani MY, Mahdy MM, Al Zuhair AA, Altamimi MS, Alshammari SN, Alshammari NM, Aowisy MAA, Alzabni WM. Evaluation of the impact of a family physician-led lifestyle clinic on overweight and obesity: A clustered randomized trial in Hail, Saudi Arabia. J Family Med Prim Care. 2025 May;14(5):2018-2025. doi: 10.4103/jfmpc.jfmpc_1969_24. Epub 2025 May 31. PMID 40547737